CLINICAL TRIAL: NCT03550170
Title: Comparing the Effectiveness of Fatigue Management Programs for People With MS
Brief Title: Fatigue Management Programs for People With MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Illinois at Chicago (Other); University of Minnesota (Other); Queen's University, Kingston, Ontario (Other); Dalhousie University (Other); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Matthew Plow, Assistant Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS-1610-37015
Record Dates: First submitted 2018-05-24; First posted 2018-06-08 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
Keywords: Fatigue; Wellness; Multiple Sclerosis; Quality of life
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Patient Portals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Teleconference (Active Comparator): Teleconference Intervention arm
  Interventions: Behavioral: Teleconference
- Internet (Active Comparator): Internet Intervention arm
  Interventions: Behavioral: Internet
- I-to-1, in-person or videoconference (Active Comparator): 1-to-1, in-person or videoconference intervention arm
  Interventions: Behavioral: 1-to-1, in-person or videoconference

INTERVENTIONS:
Behavioral: Teleconference — This intervention arm will be a 6-week, group-based course involving weekly 80-min teleconference sessions. It will be delivered in small groups (6-12 participants) to maximize participants' opportunities for interaction. A program manual divided into 6 sections, 1 for each week that includes worksheets and homework activities will be given to the participants. Occupational therapists will facilitate the sessions. Participants and the OT will dial into 1-800 conference call line on the designated date and time.
  Arms: Teleconference
Behavioral: Internet — The internet course is similar to the teleconference format. It will occur in a 6-week period and be group based; i.e., 8-12 participants will begin the intervention at the same time and interact with each other during the 6-week period. Participants will be given a username and a password to view a different session each week at a time convenient for them. Each session will include completing practice activities and sharing information (e.g., offering advice and support to one another through the discussion forum). OTs will facilitate the discussions by responding to entries, asking questions, and providing encouragement to complete sessions.
  Arms: Internet
Behavioral: 1-to-1, in-person or videoconference — Unlike the teleconference and internet courses, the number and length of sessions for the 1-to-1, in-person or videoconference course will vary over the 6-week period. The OT will cover all 6 topics, but the pace will be tailored to the participants' needs and preferences. Thus, although the topics are consistent, OTs are able to spend more time on topics that participants find pertinent to their situations. The participant and OT will be instructed to meet at least 3 times with at least 7 days between each session.
  Arms: I-to-1, in-person or videoconference

SUMMARY:
This is a multi-site randomized clinical trial comparing 3 modes of delivering the Managing Fatigue course for reducing fatigue in individuals with multiple sclerosis (MS). The primary hypothesis is that the teleconference and internet versions of the course will be noninferior to the one-on-one, in person version in terms of the primary outcome of fatigue and secondary outcome of quality of life.

DETAILED DESCRIPTION:
Fatigue is one of the most common and debilitating symptoms of multiple sclerosis (MS). MS fatigue can impact all aspects of quality of life, including physical, mental, and social function. MS fatigue is a profound barrier to participating in meaningful activities, such as employment and hobbies. Currently, the FDA has not approved medications for MS fatigue in the United States (US). However, there are empirically tested, non-pharmacological strategies that can support people with MS in reducing the impact of fatigue. Thus, the aim of the study is to compare 3 modes of delivering the Managing Fatigue course-2 telerehabilitation formats (teleconference and internet) and 1-to-1, in-person format (traditional mode of clinical service delivery)-upon outcomes important to people with MS, i.e., fatigue and its impact on physical, mental, and social function. The intervention arms will focus on reducing fatigue as a strategy to directly improve physical, mental and social functioning.

ELIGIBILITY:
Inclusion Criteria:

* Self-report diagnosis of MS
* Age ≥ 18 years
* Fatigue Severity Scale score ≥ 4
* Ability to speak English

Exclusion Criteria:

* Individual must be capable of providing consent (Assessed with questionnaire)
* Unable to access the internet or unable to travel to in-person sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Plow, PhD, Principal Investigator — Case Western Reserve University
Locations (3):
- United States (3):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Case Western Reserve University, Cleveland, Ohio

REFERENCES:
- [Derived] Plow M, Packer T, Mathiowetz VG, Preissner K, Ghahari S, Sattar A, Bethoux F, Finlayson M. REFRESH protocol: a non-inferiority randomised clinical trial comparing internet and teleconference to in-person 'Managing Fatigue' interventions on the impact of fatigue among persons with multiple sclerosis. BMJ Open. 2020 Aug 16;10(8):e035470. doi: 10.1136/bmjopen-2019-035470. PMID 32801193

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled participants would only be excluded from the study before assignment to groups if they did not meet the inclusion criteria stated in the protocol.
Groups:
- One-to-One: One-to-one intervention arm: Unlike the teleconference and internet courses, the number and length of sessions for the one-to-one course will vary over the 6-week period. The OT will cover all 6 topics, but the pace will be tailored to the participants' needs and preferences. Thus, although the topics are consistent, OTs are able to spend more time on topics that participants find pertinent to their situations. The participant and OT will be instructed to meet at least 3 times with at least 7 days between each session.
Period: Overall Study
Arm/Group | Teleconference | Internet | One-to-One
Started | 196 | 197 | 197
Completed | 174 | 186 | 172
Not Completed | 22 | 11 | 25

BASELINE CHARACTERISTICS:
Groups:
- One-to-One: One-to-One intervention arm
  One-to-one: Unlike the teleconference and internet courses, the number and length of sessions for the 1-to-1, in-person or videoconference course will vary over the 6-week period. The OT will cover all 6 topics, but the pace will be tailored to the participants' needs and preferences. Thus, although the topics are consistent, OTs are able to spend more time on topics that participants find pertinent to their situations. The participant and OT will be instructed to meet at least 3 times with at least 7 days between each session.
- Total: Total of all reporting groups
Arm/Group | Teleconference | Internet | One-to-One | Total
Number analyzed (Participants) | 196 | 197 | 197 | 590
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (11) | 53 (11) | 51 (12) | 52 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 158 | 161 | 485
  Male | 30 | 39 | 36 | 105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 4 | 8 | 9 | 21
  Non-Hispanic | 191 | 188 | 187 | 566
  African American | 24 | 23 | 23 | 70
  Asian | 1 | 1 | 0 | 2
  White | 165 | 166 | 171 | 502
  American Indian/Alaska Native | 0 | 0 | 0 | 0
  Hawaiian/Pacific Islander | 0 | 0 | 0 | 0
  Multiracial | 6 | 3 | 3 | 12
  Missing Race | 0 | 4 | 0 | 4
Fatigue Impact Scale [Mean (Standard Deviation); unit: units on a scale] | 68.62 (33.78) | 67.73 (33.03) | 68.10 (33.61) | 68.15 (33.42)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fatigue Levels
Description: Fatigue will be assessed with Fatigue Impact Scale. Fatigue Impact Scale is a 40-item questionnaire that measures impact of fatigue on day-to-day life. Scale ranges from "no problem" (0) to "extreme problem" (4). Total scores will be computed by summing responses for each item. Scores can range from 0 to 160 with a higher score indicating worse fatigue.
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- One-to-one: One-to-one intervention arm
  One-to-one, in-person or videoconference: Unlike the teleconference and internet courses, the number and length of sessions for the 1-to-1, in-person course will vary over the 6-week period. The OT will cover all 6 topics, but the pace will be tailored to the participants' needs and preferences. Thus, although the topics are consistent, OTs are able to spend more time on topics that participants find pertinent to their situations. The participant and OT will be instructed to meet at least 3 times with at least 7 days between each session.
Arm/Group | Teleconference | Internet | One-to-one
Number analyzed (Participants) | 196 | 197 | 197
score on a scale | 50.98 (2.08) | 56.88 (0.59) | 57.87 (1.34)
Statistical Analysis 1: Comparison: Teleconference vs One-to-one; A generalized estimating equation (GEE) served as the primary analysis tool for modeling the longitudinal scores of the primary outcome - Fatigue Impact Scale (FIS); Test type: Non-Inferiority — Non-inferiority was established using the prespecified margin of inferiority of 10 points on the total composite score of the Fatigue Impact Scale; Slope = 4.89, 90% CI 2-sided [0.67 to 9.11], Standard Error of Mean 2.57 — Comparison of teleconference to one-to-one at 6 months
Statistical Analysis 2: Comparison: Internet vs One-to-one; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Slope = 6.12, 90% CI 2-sided [0.98 to 11.26], Standard Error of Mean 2.62 — Comparison of internet to one-to-one at 6 months

2. Secondary Outcome: Change From Baseline in Health-related Quality of Life: Psychological Composite
Description: Multiple Sclerosis Impact Scale (MSIS) was used to measure health-related quality of life. It consists of 29 self-report questions. The psychological composite score is calculated on a scale between 1 and 100. Higher scores indicate worse health-related quality of life.
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teleconference | Internet | One-to-One
Number analyzed (Participants) | 163 | 131 | 145
score on a scale | 40.93 (23.05) | 38.66 (21.80) | 37.77 (21.68)
Statistical Analysis 1: Comparison: Teleconference vs Internet vs One-to-One; Test type: Superiority; p = 0.10, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the course of data collection for each participant, which was 6 months long.
Groups:
- One-to-One: One-to-one intervention arm
  1-to-1: Unlike the teleconference and internet courses, the number and length of sessions for the 1-to-1, in-person course will vary over the 6-week period. The OT will cover all 6 topics, but the pace will be tailored to the participants' needs and preferences. Thus, although the topics are consistent, OTs are able to spend more time on topics that participants find pertinent to their situations. The participant and OT will be instructed to meet at least 3 times with at least 7 days between each session.
Arm/Group | Teleconference | Internet | One-to-One
All-Cause Mortality (participants affected / at risk) | 0/196 | 0/197 | 0/197
Serious Adverse Events (participants affected / at risk) | 0/196 | 0/197 | 0/197
Other Adverse Events (participants affected / at risk) | 0/196 | 0/197 | 0/197

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT03550170/Prot_SAP_000.pdf